CLINICAL TRIAL: NCT06300762
Title: A Prospective, Multicenter, Partially Assessor Blinded, Randomised, Open Label, Parallel, Comparative Clinical Trial to Evaluate the Exudate Management Performance of Cutimed Sorbion Product Range
Brief Title: RCT Exudate Management Cutimed Sorbion Product Range
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BSN Medical GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C3079
Record Dates: First submitted 2024-02-20; First posted 2024-03-08 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Two assessors are blinded to evaluate some outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cutimed Sorbion products (Experimental): Within this arm the Cutimed Sorbion (Cutimed® Sorbion® Sachet/Sana/Border) products will be used for exudate managment.
  Interventions: Device: Superabsorbent dressing application
- Zetuvit (RespoSorb) products (Active Comparator): Within this arm the comperator products Zetuvit® Plus/(RespoSorb® Super), Zetuvit® Plus Silicone/(RespoSorb® Silicone) and Zetuvit® Plus Silicone Border/(RespoSorb® Silicone Border) will be used for exudate management.
  Interventions: Device: Superabsorbent dressing application

INTERVENTIONS:
Device: Superabsorbent dressing application — Cutimed Sorbion or Zetuvit plus (RespoSorb) application to maintain wound exudate

SUMMARY:
The fluid handling capacity of superabsorbent dressings varies depending on the design and construction. The use of effective advanced wound dressings is a promising strategy to achieve adequate absorption of wound exudate and malodour promoting wound healing. The aim of the current study is to determine whether there is a difference in the clinical performance of exudate absorption with two commonly used CE-marked superabsorbent dressings when used on VLUs in routine wound care.

As primary objective the dressing´s absorption performance and its ability to prevent skin maceration and leakage of the wound dressing will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is informed about the trial, understands the nature of the study and provides written informed consent prior to study enrolment
2. Participant is mentally and physically able to participate in this study
3. Men, women, diverse ≥ 18 years
4. Participant complies with study visit schedule
5. Participant agrees to comply with all standard therapies (e.g., with regards to compression therapy)
6. Participant suffers from lower leg ulcer* (including the ankle but not the feet) indicated to be treated with the study deviceinvestigational devices, requiring compression and fulfilling the following:
7. Ulcer is not younger than 4 weeks and not older than 1 year
8. Ulcer is ranging between 2 cm2 and 800 cm2
9. One side of the ulcer is not extending 40 cm
10. Depth of ulcer < 2 cm
11. Ankle-brachial pressure index (ABPI) of >0.8 and ≤1.3, measurement not older than 12 months * Participants with more than one ulcer are eligible for inclusion, however only one ulcer per patient will be included in the study.

Exclusion Criteria:

1. Participant already participates in this study with one ulcer (only one ulcer per participant is allowed)
2. Participant is expected not to be willing or able to follow the study outlines and requirements
3. Participant suffers from systemic infectious disease(s) known to negatively influence wound healing, such as AIDS
4. Participant is undergoing an immuno-compromising therapy, such as systemic antineoplastic drugs and/or systemic corticosteroids
5. Participant uses any medication that could potentially delay the wound healing ability
6. Participant is an employee (staff or student) of the hospital site (institute) or the sponsor or is in a dependent relationship with a member of site or sponsor staff, e.g. child, spouse etc.
7. Participant is pregnant or currently breastfeeding
8. Participant reporting (and/or suspected by investigator) addiction from alcohol or drugs or is substituted e.g., by Methadone

8. Participant suffers from alcohol or drug addiction or is substituted e.g., by Methadone 9. Participant is or has been included in another clinical investigation with medical devices or pharmaceutical drugs at present or during the past 30 days 10. Participant with a history of sensitivity to any of the components of the study product 11. Participant whose leg ulcers are clinically infected (e.g., erysipelas) or malignant 12. Study ulcer requiring negative pressure wound therapy or hyperbaric oxygen during the trial 13. The ulcer has exposed bone, tendon, ligaments and/or joint 14. History of radiation at the study ulcer site 15. Participant's lesion is a primary skin cancer 16. Participant's lesion is the manifestation of a metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2024-08-10 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Exudate management performance | up to 30 days
  Capability to main exudate uptake and retention as well as leakage prevention

SECONDARY OUTCOMES:
Dressing change frequency | up to 30 days
  Number of required intermediate dressing changes between study visits and assessement fo reasons for
Moisture-associated skin damages | up to 30 days
  Occurrence of moisture-associated skin damages
Occurrence clinical relevant peri-wound skin changes | up to 30 days
  Effect of product use on peri-wound skin such as reddening, swelling, clinical relevant skin detoriations
Changes in wound tissue and general wound pain | up to 30 days
  Effect of product use on the wound considering wound tissue and slough on the wound as well as the general wound pain assessed using a 11 visual analogue scale from 0-10 (0= not pain, 10=most imaginable pain for the participant)
Need for debridement after product removal | up to 30 days
  Evaluation of the soft debridement effect of Cutimed Sorbion products during dressing removal: is the soft debrimdent supporting wound cleansing and eases addtional wound debridement
Patient satisfaction with treatment and product | final study visit
  Patient´s impressions about treatment and felt protection for leakage when using the product and assessment of individually felt wearing comfort
HCP satisfaction with treatment and product | final study visit
  HCP´s satisfaction with treatment and product performance to manage wound exudate, check if treatment need have been met be the product
Changes in quality of life using the "Wound-QoL 14" (short questionnaire measuring quality of life in patients with chronic wounds based on three established disease-specific instruments) | day 0 and day 30
  Fourteen items are scored using a Likert-type scale as either 'not at all', 'a little', 'moderately', 'quite a lot' or 'very much'. Item data are calculated building a global score and the 3 subscores "Body", "Psyche/Well-being" and the "Everyday life". In increase in quality of life is indicated by decreasing sub- and/or global score.

CONTACTS AND LOCATIONS:
Locations (3):
- Niels Stensen Klinik, Christliches-Klinikum-Melle, Melle, Niedersachsten, Germany
- United Kingdom (2):
  - Mid Yorkshire Teaching NHS Trust Pinderfields Hospital, Wakefield, West Yorkshire
  - Northumbria Healthcare NHS Foundation Trust, Ashington

IPD SHARING:
Plan to Share IPD: No